CLINICAL TRIAL: NCT00025428
Title: Treatment Of Children Over The Age Of 1 Year With Unresectable Localized Neuroblastoma Without MYCN Amplification
Brief Title: Combination Chemotherapy Before Surgery in Treating Children With Localized Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Collaborators: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068960; SIOP-NB-2009; CCLG-NB-2000-09; EU-20107
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Neuroblastoma
Keywords: localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase III trial to determine the effectiveness of combination chemotherapy given before surgery in treating children who have localized neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the outcome, in terms of local control, event-free survival, and overall survival, of children with localized unresectable neuroblastoma without MYCN amplification treated with carboplatin, etoposide, cyclophosphamide, doxorubicin, and vincristine followed by surgery.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV over 1 hour and etoposide IV over 2 hours on days 1-3 (courses 1 and 3). Patients receive cyclophosphamide IV over 1 hour on days 1-5 (or orally on days 2 and 3), doxorubicin IV over 6 hours on days 4-5, and vincristine IV on days 1 and 5 (courses 2 and 4). Treatment repeats every 21 days for 4 courses. Patients then undergo surgical resection followed by 2 additional courses of chemotherapy.

Patients are followed at months 8, 10, 12, 16, 20, 24, 30, 36, 42, 48, and 60.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized unresectable neuroblastoma

  * Stage II or III
  * No MYCN amplification

PATIENT CHARACTERISTICS:

Age:

* Over 1

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-12; Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Event-free survival at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Janice A. Kohler, MD, FRCP, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (12):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Odense University Hospital, Odense, Denmark
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Children's Hospital, Cologne, Germany
- Istituto Giannina Gaslini, Genoa, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Hospital Universitario LA FE, Valencia, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Southampton University Hospital NHS Trust, Southampton, England, United Kingdom